CLINICAL TRIAL: NCT00219440
Title: A Portion-controlled Diet Will Prevent Weight Gain in Diabetics Treated With ACTOS
Acronym: TAKE II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, George A. Bray, Professor, Adjunct, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 24005
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): ACTOS plus standard diet
  Interventions: Other: Actos plus standard diet
- B (Experimental): Actos plus structured diet
  Interventions: Other: Actos plus structured diet
- C (Experimental): Metformin plus standard diet
  Interventions: Other: Metformin plus standard diet

INTERVENTIONS:
Other: Actos plus standard diet — Actos plus standard diet
  Arms: A
Other: Actos plus structured diet — Actos plus structured diet
  Arms: B
Other: Metformin plus standard diet — Metformin plus standard diet
  Arms: C

SUMMARY:
We hypothesized that a portion controlled diet would prevent the weight gain associated with the use of a peroxisome profliferator-activated receptor-gamma (PPAR-g). This is a 4 months randomized clinical trial in type 2 diabetics who are treated with pioglitazone and a standard diet, pioglitazone and a portion-controlled diet and metformin with a standard diet.

DETAILED DESCRIPTION:
A total of 60 male and female type 2 diabetic subjects will be recruited and randomized into 1 of 3 treatment groups for the 4 months long trial

1. ACTOS plus a standard diet
2. ACTOS plus a portion-controlled diet
3. Metformin plus a standard diet. The end-point of the trial is the change in body fat content from baseline to the end of the trial

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 35 to 75 who have type 2 diabetes mellitus

Exclusion Criteria:

* Individuals with co-existing other diseases

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2003-02; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
glucose | 4 months

SECONDARY OUTCOMES:
Change in lipids | 4 months
blood pressure | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: George A Bray, MD, Principal Investigator — Pennington Center
Locations (1):
- Pennington Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Martin CK, Gupta AK, Smith SR, Greenway FL, Han H, Bray GA. Effect of pioglitazone on energy intake and ghrelin in diabetic patients. Diabetes Care. 2010 Apr;33(4):742-4. doi: 10.2337/dc09-1600. Epub 2010 Jan 12. PMID 20067964
- [Derived] Gupta AK, Smith SR, Greenway FL, Bray GA. Pioglitazone treatment in type 2 diabetes mellitus when combined with portion control diet modifies the metabolic syndrome. Diabetes Obes Metab. 2009 Apr;11(4):330-7. doi: 10.1111/j.1463-1326.2008.00965.x. PMID 19267711